CLINICAL TRIAL: NCT06641024
Title: Phase I Clinical Study of CD19-targeting Chimeric Antigen Receptor T Lymphocyte (MC-1-50) for the Treatment of Relapsed/Refractory CD19-positive B-cell Acute Lymphoblastic Leukemia (B-ALL)
Brief Title: Clinical Research of CD19 Targeted CAR-T Cell in Relapsed/ Refractory B-ALL
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB12
Record Dates: First submitted 2024-09-27; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Acute Lymphoblastic Leukemia, in Relapse; Refractory Acute Lymphoblastic Leukemia
Keywords: B-ALL; CAR-T
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MC-1-50 (Experimental): Patients will be be treated with CD19 CAR- T cells
  Interventions: Biological: MC-1-50

INTERVENTIONS:
Biological: MC-1-50 — A single infusion of CD19 CAR-T cells will be administered intravenously after lymphodepletion chemotherapy

SUMMARY:
This is a single-arm, open-label, dose-escalation phase I clinical study to explore the safety, tolerability, and cytokinetic characteristics of MC-1-50 cell formulation, and to preliminarily observe the efficacy of MC-1-50 cell formulation in subjects with relapsed/refractory CD19-positive B Cell Acute Lymphoblastic Leukemia.

DETAILED DESCRIPTION:
Based on the specific CD19-targeting CAR-T developed on the PrimeCARTM platform, the cell preparation time is about 3 days, which can greatly shorten the waiting time of patients, improve production efficiency and reduce production costs. At the same time, MC-1-50 products have a high proportion of T naive cells, which can play a therapeutic effect at a very low infusion dose to improve safety. In this study, a "3+3" design was adopted, and three dose groups were set up with 1×10^5/kg, 3×10^5/kg, and 5×10^5/kg CAR-positive cells, respectively (the upper limit of the total number of cells was not more than 5×10^7 CAR-positive cells). All subjects received only one infusion of MC-1-50 cells.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or their guardian agrees to participate in this clinical trial and sign the ICF, indicating their understanding of the purpose and procedures of this clinical trial and willingness to participate in the study;
2. Age ≥ 18 years old (including threshold), gender not limited;
3. Diagnosed with B-cell acute lymphoblastic leukemia and meeting one of the following conditions:

   1. Refractory B-ALL: Early refractory patients who have not achieved complete remission of bone marrow after two courses of first-line systemic therapy upon initial diagnosis;
   2. Relapsed B-ALL:

      ① Early relapsed after complete remission (< 12 months);

      ② Late relapsed after complete remission (≥ 12 months) requires systemic therapy again, but if complete remission is not achieved or early treatment response is poor;

      ③ Having experienced 2 or more times bone marrow relapse;

      ④ Relapsed after allogeneic hematopoietic stem cell transplantation;
   3. Individuals with Philadelphia chromosome positive (Ph+) disease are eligible if they have relapsed/refractory disease despite treatment with at least 2 different tyrosine kinase inhibitors (TKIs); (Note: Except for those who are intolerant to TKI therapy, or have T315i mutations);
4. Flow cytometry confirms the expression of CD19 in leukemia cells in the bone marrow. In individuals previously treated with targeted CD19 antibodies (such as blinatumomab), the proportion of CD19 positive cells in leukemia cells must be ≥ 90%;
5. Morphological disease in the bone marrow (≥ 5% blasts);
6. ECOG score 0-1;
7. Expected survival time of more than 12 weeks;
8. Adequate renal, hepatic, pulmonary and cardiac function defined as:

   1. Cardiac function: Echocardiography indicates left ventricular ejection fraction ≥ 50%;
   2. Renal function: serum creatinine ≤ 2.0 × ULN, or creatinine clearance rate ≥ 60ml/min (Cockcroft Gault formula);
   3. Hepatic function: ALT and AST ≤ 3.0 × ULN (may be relaxed to ≤ 5.0 × ULN in cases of combined liver infiltration);
   4. Total bilirubin ≤ 2.0 × ULN (Gilbert syndrome requires total bilirubin ≤ 3.0 × ULN);
   5. Pulmonary function: Blood oxygen saturation is ≥ 92% in non oxygen state.
9. No serious mental disorders;
10. Meet standards for apheresis or venous blood collection, and no other cell collection contraindications;
11. Women of childbearing age who have a negative blood pregnancy test and all subjects agree to use reliable and effective contraceptive methods (excluding safe period contraception) for contraception within one year after receiving MC-1-50 cell infusion from the time of signing the informed consent form. Including but not limited to: abstinence, implantable progestogen contraceptives that can inhibit ovulation; Intrauterine device (IUD); Intrauterine hormone release system; Spouse vasectomy; Compound hormone contraceptives that can inhibit ovulation (oral, vaginal, and transdermal); Progesterone contraceptives (oral or injectable) that can inhibit ovulation; When male subjects have sex with fertile women, they must agree to use barrier contraception (such as condom plus spermicidal foam/gel/film/emulsion/suppository). At the same time, participants should commit not to donate eggs (oocytes, oocytes) or sperm for assisted reproduction within one year after cell infusion.

Exclusion Criteria:

1. Isolated extramedullary disease;
2. Central nervous system abnormalities: defined as CNS-2 and 3 according to NCCN guidelines (note: CNS-2 and 3 can be screened, but must be treated and recovered to CNS-1 before lymphodepleting chemotherapy and infusion);
3. Transformation of chronic myeloid leukemia to acute biphenotypic leukemia;
4. Individuals who have received CAR-T therapy or other gene modified cell therapies;
5. Prior to apheresis, the following anti-tumor treatments have been received: chemotherapy, targeted therapy, and other drug treatments within 14 days or at least 5 half lives (whichever is shorter); Received radiation therapy within 14 days;
6. HBsAg or HBcAb positive and HBV DNA is greater than the normal range; HCV antibody is positive and HCV RNA greater than the normal range; HIV antibody positive; syphilis positive; CMV DNA positive;HBsAg or HBcAb positive and HBV DNA is greater than the normal range; HCV antibody is positive and HCV RNA greater than the normal range; HIV antibody positive; syphilis positive;
7. Suffered from any of the following heart diseases:

   1. New York Heart Association (NYHA) stage III or IV congestive heart failure;
   2. Within the 6 months prior to enrollment, there has been a myocardial infarction, or a coronary artery bypass grafting (CABG) or stent implantation surgery has been performed;
   3. History of ventricular arrhythmias requiring treatment or unexplained syncope (excluding cases caused by vasovagal or dehydration);
   4. History of severe non-ischemic cardiomyopathy;
8. Uncontrollable infection in the 2 weeks before enrollment;
9. Acute grade 2-4 graft-versus-host disease (GVHD) or moderate to severe chronic GVHD within the first 4 weeks of enrollment;
10. If a cerebrovascular accident or seizure occurs within the first 6 months of enrollment;
11. Active autoimmune diseases;
12. Deep vein or deep artery embolism event within the past 6 months prior to enrollment;
13. Poor control of hypertension during screening is defined as systolic blood pressure ≥ 160mmHg and/or diastolic blood pressure ≥ 100mmHg (blood pressure values are measured based on the average of three readings taken at least 2 minutes apart. Patients with blood pressure ≥ 160/100mmHg at the initial screening can receive antihypertensive treatment, and if good control is achieved after treatment and blood pressure<160/100mmHg, enrollment can be performed);
14. History of malignancy other than fully treated cervical carcinoma in situ, basal cell or squamous cell carcinoma of the skin, local prostate cancer after radical surgery, and ductal carcinoma in situ of the breast after radical surgery;
15. (attenuated) Live vaccine ≤ 4 weeks prior to enrollment;
16. Have participated in other clinical trials within one month or five drug half lives (whichever is shorter) before enrollment;
17. Women who are pregnant or breastfeeding, and male or female subjects who plan to have children within 1 year after receiving MC-1-50 cell infusion;
18. Other situations considered by the investigator to be unsuitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2039-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 1 month
  Dose-limiting toxicity after CD19 CAR-T cell infusion
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 1 month
  The incidence of adverse events after CAR-T cell infusion was assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, version 5.0)

SECONDARY OUTCOMES:
AUCS of MC-1-50 cells [Cell dynamics] | 3 months
  AUCS is defined as the area under the curve in 90 days
CMAX of MC-1-50 cell preparation [Cell dynamics] | 3 months
  CMAX is defined as the highest concentration of MC-1-50 cells expanded in peripheral blood
TMAX of MC-1-50 cell preparation[Cell dynamics] | 3 months
  TMAX is defined as the time to reach the highest concentration
Pharmacodynamics of MC-1-50 cell preparation[Cell dynamics] | 3 months
  The clearance degree of CD19-positive B cells in peripheral blood was detected by flow cytometry at the visit points specified in the research protocol
Immunogenicity of pCAR-19B cells | 3 months
  The anti-CAR antibody was detected by ELISAt the visit points specified in the research protocol
Objective response rate after MC-1-50 infusion [Efficacy] | 3 months
  Objective response rate after pCAR-19B infusion [Efficacy]

OTHER OUTCOMES:
Objective response rate after MC-1-50 infusion [Long-term Efficacy] | 2 years
  Objective response rate includes CR, CRi
Duration of Response (DOR) after MC-1-50 infusion [Long-term Efficacy] | 2 years
  DOR will be assessed from the first assessment of CR/PR to the first assessment of recurrence or progression of the disease or death from any cause
Progress-free survival(PFS) after MC-1-50 infusion [Long-term Efficacy] | 2 years
  PFS will be assessed from the first MC-1-50 cell infusion to death from any cause or the first assessment of progression
Event-Free survival(EFS) after MC-1-50 infusion [Long-term Efficacy] | 2 years
  EFS will be assessed from the first MC-1-50 cell infusion to death from any cause or Disease progression or Treatment failure
Overall survival(OS) after MC-1-50 infusion [Long-term Efficacy] | 2 years
  OS will be assessed from the first MC-1-50 cell infusion to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Rui Jin hospital, Shanghai Jiao Tong university school of medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No